CLINICAL TRIAL: NCT01401751
Title: Feasibility Study Assessing The Ability Of An Insulin Pump-Controlling Algorithm To Minimize Hypoglycemia And Hyperglycemia In Patients With Type 1 Diabetes In A Clinical Research Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Animas Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 3076823
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Other): non-randomized, uncontrolled, feasibility study
  Interventions: Device: Hypoglycemia-Hyperglycemia Minimizer System

INTERVENTIONS:
Device: Hypoglycemia-Hyperglycemia Minimizer System — Hypoglycemia-Hyperglycemia Minimizer System, consisting of an subcutaneous insulin infusion pump, subcutaneous continuous glucose monitoring system, and a controller algorithm

SUMMARY:
The purpose of this study is to evaluate the performance of an insulin pump controlling algorithm while the subject is under close medical supervision in the Clinical Research Center (CRC) setting.

DETAILED DESCRIPTION:
This study is a non-randomized, uncontrolled feasibility study that looks to enroll people with type 1 diabetes who are currently using an insulin pump. During the subject's participation, the study staff will closely monitor the study subject in a clinical research center environment for approximately 24 hours, while controller algorithm determined insulin doses are delivered by an insulin pump, and utilizing continuous glucose monitoring results.

Total subject participation approximately 1 week for screening to completion. This includes approximately 24 hours usage of the investigation device in the clinical research center under close medical supervision.

ELIGIBILITY:
Summary of Key inclusion/exclusion criteria:

Inclusion Criteria:

* Age 21-65 years
* Type 1 diabetes mellitus for at least one year
* Using an insulin infusion pump for at least the past 6 months

Exclusion Criteria:

* Pregnancy
* History of diabetic ketoacidosis (DKA) in the past six months
* History of severe hypoglycemia (seizure, unconsciousness) in the past 6 months

Other Inclusion/Exclusion criteria apply.

Please contact clinical study site for complete details.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2011-12-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of the System while the subject is under close medical supervision in the Clinical Research Center (CRC) setting. | End of Study - in approximately 5 months from first subject enrolled
  Measuring the response of the investigational device, including insulin delivery dosing changes in response to glucose changes. Also, the ability of the system to mitigate Hypoglycemia.

SECONDARY OUTCOMES:
Safety Evaluation | End of Study - in approximately 5 months from first subject enrolled
  Measuring the following:
  * the number and type of adverse events, including Adverse device effects, Serious Adverse Events, Unanticipated Adverse Device Effects, device malfunctions
  * Resulting glucose data from 24 hour clinical research center visit

CONTACTS AND LOCATIONS:
Overall Officials: Howard Zisser, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States